CLINICAL TRIAL: NCT05328401
Title: To Evaluate the Therapeutic Effect of Laser Acupuncture in Patients with Acute or Subacute Post Stroke Shoulder Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202200086A3; 202200086A3C502 (Other: ChangGungMH)
Record Dates: First submitted 2022-03-22; First posted 2022-04-14 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Post Stroke Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (verum laser acupuncture group ) (Experimental): After blind random allocation, investigators applied verum laser acupuncture on patient with shoulder pain after stroke.
  Interventions: Device: Verum laser acupuncture
- Control group (sham laser acupuncture group) (Sham Comparator): After blind random allocation, investigators applied sham laser acupuncture on patient with shoulder pain after stroke.
  Interventions: Device: Sham laser acupuncture

INTERVENTIONS:
Device: Verum laser acupuncture — Applied verum laser acupuncture on specific acupoints in patient with post stroke shoulder pain.
  Arms: Intervention group (verum laser acupuncture group )
Device: Sham laser acupuncture — Applied sham laser acupuncture on specific acupoints in patient with post stroke shoulder pain.
  Arms: Control group (sham laser acupuncture group)

SUMMARY:
Investigators propose a research design protocol to evaluate the efficacy of laser acupuncture in improving shoulder pain and improving shoulder function recovery after stroke.

DETAILED DESCRIPTION:
Shoulder pain after stroke, also known as hemiplegic shoulder pain, is one of the common complications after stroke. The overall incidence rate increases with the time after stroke.The existing treatment methods for shoulder pain after stroke are divided into non-drug and drug. Investigators propose a research design protocol to evaluate the efficacy of laser acupuncture in improving shoulder pain and improving shoulder function recovery after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Beyond the age of 20.
* Normal consciousness before and after stroke who can reply and fill in the questionnaire.
* Subacute (subacute phase: 7 days to 6 months after stroke) and Chronic (chronic phase: more than 6 months after stroke) with shoulder pain after stroke and in post- stroke recovery period.
* Stop taking painkillers for more than 1 day,
* Without received intramuscular drugs (steroids, botulinum toxin, glucose, etc.) injections in the shoulder joint or around the shoulder for more than 2 weeks
* Those willing to sign the written subject consent form.

Exclusion Criteria:

* Participants with shoulder pain symptoms before the stroke
* Acute shoulder trauma on the affected side of shoulder pain in the past.
* Surgery on the affected side of shoulder pain in the past.
* Those who cannot complete the scale assessment due to aphasia, post-stroke depression, and obvious cognitive impairment.
* Women who are pregnant or planning to become pregnant.
* Those who have a history of epilepsy and are receiving anti-epileptic drug treatment.
* Who are receiving any herbal or folk remedies related to shoulder pain.
* Any other conditions deemed unsuitable in the assessment of the responsible physician.
* Those who have not signed the written subject consent form.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-04-16 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Passive range of motion of shoulder | 3 weeks
  Measuring the passive range of motion (Scale unit: angular degree) of shoulder (Abduction ranged from 0-180 degree, flexion ranged from 0-180 degree, external rotation ranged from 0-90 degree) of patient with shoulder pain. The higher degree of range of motion mean the better outcome.
Numerical rating scale | 3 weeks
  Measuring the pain level by Numerical rating scale (scale unit: point). The scales ranged form 1 to 10 and the higher scores mean the worse outcome.

SECONDARY OUTCOMES:
Brief Pain Inventory - Short Form (BPI-sf) | 3 weeks
  Measuring the level of daily life effect by shoulder pain by Visual graphic rating scale (scale unit: point) of BPI-sf. The scales ranged form 1 to 10 and the higher scores mean the worse outcome.
Visual graphic rating scale (VGRS) of ShoulderQ | 3 weeks
  Measuring the pain level on deferent time points by Visual graphic rating scale (scale unit: point) of ShoulderQ. The scales ranged form 1 to 10 and the higher scores mean the worse outcome.
Meridian energy by Meridian Energy Analysis Devices | 3 weeks
  Meridian Energy Analysis Devices (MEADs) is a non-invasive meridian energy measurement tool used to Measure the meridian energy of patient. By measuring the current value (scale unit: micro ampere, uA) in the subject's limbs, investigators estimate the energy meridian energy. The higher the current energy value, the higher the meridian energy.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Wei Chang, Study Director — Chang Gung Medical Foundation
Locations (1):
- Chang Gung Memorial Hospital, Keelung Medical Center, Keelung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
We do not share the data of this study.